CLINICAL TRIAL: NCT02405442
Title: A Phase 2, Double-blind, Randomized, Placebo-Controlled, Multicenter Study Evaluating the Safety and Efficacy of GS-5745 in Subjects With Moderately to Severely Active Crohn's Disease
Brief Title: Safety and Efficacy of Andecaliximab in Participants With Moderately to Severely Active Crohn's Disease
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GS-US-395-1663; 2015-001249-10 (EudraCT Number)
Record Dates: First submitted 2015-03-27; First posted 2015-04-01 (Estimated); Results first posted 2019-03-28 (Actual); Last update posted 2019-04-23 (Actual); Status verified 2019-04

CONDITIONS: Crohn's Disease
MeSH Terms: conditions — Crohn Disease | interventions — andecaliximab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Andecaliximab 150 mg Every 2 Weeks (Experimental): Double-Blind Phase: Participants will receive 1 single-use prefilled syringe (PFS) of andecaliximab 150 mg and matching placebo coadministered at Weeks 0, 2, 4, and 6 and 2 single-use PFS of placebo coadministered at Weeks 1, 3, 5, and 7. Open-Label Phase: Participants will be eligible to enroll in the Open-Label Phase to receive andecaliximab 150 mg weekly for an additional 44 weeks. Extended Treatment Phase: Participants who complete Week 52 assessments will be eligible to enter into the Extended Treatment Phase to continue treatment with andecaliximab 150 mg for an additional 156 weeks.
  Interventions: Drug: Andecaliximab; Drug: Placebo
- Andecaliximab 150 mg Weekly (Experimental): Double-Blind Phase: Participants will receive 1 single-use PFS of andecaliximab 150 mg and matching placebo coadministered weekly for 8 weeks. Open-Label Phase: Participants will be eligible to enroll in the Open-Label Phase to receive andecaliximab 150 mg weekly for an additional 44 weeks. Extended Treatment Phase: Participants who complete Week 52 assessments will be eligible to enter into the Extended Treatment Phase to continue treatment with andecaliximab 150 mg for an additional 156 weeks.
  Interventions: Drug: Andecaliximab; Drug: Placebo
- Andecaliximab 300 mg Weekly (Experimental): Double-Blind Phase: Participants will receive 2 single-use PFS of andecaliximab 150 mg coadministered weekly for 8 weeks. Open-Label Phase: Participants will be eligible to enroll in the Open-Label Phase to receive andecaliximab 150 mg weekly for an additional 44 weeks. Extended Treatment Phase: Participants who complete Week 52 assessments will be eligible to enter into the Extended Treatment Phase to continue treatment with andecaliximab 150 mg for an additional 156 weeks.
  Interventions: Drug: Andecaliximab
- Placebo (Placebo Comparator): Double-Blind Phase: Participants will receive 2 single-use PFS of placebo coadministered weekly for 8 weeks. Open-Label Phase: Participants will be eligible to enroll in the Open-Label Phase to receive andecaliximab 150 mg weekly for 44 weeks. Extended Treatment Phase: Participants who complete Week 52 assessments will be eligible to enter into the Extended Treatment Phase to continue treatment with andecaliximab 150 mg for an additional 156 weeks.
  Interventions: Drug: Andecaliximab; Drug: Placebo

INTERVENTIONS:
Drug: Andecaliximab — Andecaliximab administered via subcutaneous (SC) injection
  Other Names: GS-5745
Drug: Placebo — Placebo to match andecaliximab administered via SC injection
  Arms: Andecaliximab 150 mg Every 2 Weeks; Andecaliximab 150 mg Weekly; Placebo

SUMMARY:
This study will primarily evaluate the safety and efficacy of andecaliximab in adults with active Crohn's disease. The study will consist of a Double-Blind Phase of 8 weeks followed by an Open-Label Extension. Participants who complete the Double-Blind Phase will be eligible to enroll in the optional Open-Label Extension for an additional 44 weeks. Participants who complete Week 52 assessments will be eligible to enter the Extended Treatment Phase to continue treatment with andecaliximab for an additional 156 weeks.

ELIGIBILITY:
Key Inclusion Criteria:

* Ability to provide a written informed consent
* Females of childbearing potential must have a negative pregnancy test at screening and baseline
* Documented diagnosis of Crohn's disease with a minimum disease duration of 6 months with involvement of the ileum and/or colon at a minimum
* Moderately to severely active Crohn's disease as defined by a Crohn's Disease Activity Index (CDAI) total score between 220-450 (inclusive) AND with evidence of active disease as measured by ileocolonoscopy
* Within the previous 5 years, demonstrated an inadequate clinical response or intolerance of at least one of the following agents:

  * Corticosteroids
  * Immunomodulators
  * Tumor necrosis factor-alpha (TNFα) antagonists
  * Vedolizumab
* May be receiving the following drugs:

  * Oral 5-aminosalicylate (5-ASA)
  * Oral corticosteroid therapy
  * Antidiarrheals for chronic diarrhea
  * Azathioprine or 6-mercaptopurine (6-MP) or methotrexate
  * Antibiotics for the treatment of Crohn's disease
* Able to comply with the dosing instructions for study drug and able to comply with the study visits and requirements

Key Exclusion Criteria:

* Evidence of abscess at screening
* Extensive colonic resection (subtotal or total colectomy) or history of > 2 small bowel resections
* Ileostomy, colostomy, or symptomatic stenosis of the intestine
* Current use of oral corticosteroids at a dose equivalent to > 30 mg/day of prednisone
* Ulcerative colitis or indeterminate colitis
* Short bowel syndrome
* Stool sample positive for Clostridium difficile (C. difficile) toxin, E. coli, Salmonella, Shigella, Campylobacter or Yersinia
* Treatment with any monoclonal antibody within 4 weeks of screening
* History or evidence of colonic mucosal dysplasia
* HIV, hepatitis B, hepatitis C, or tuberculosis (TB) infection
* Participated in a clinical study with an investigational drug or biologic within the last 30 days
* Any chronic medical condition (including, but not limited to, cardiac or pulmonary disease) that, in the opinion of the investigator, would make the individual unsuitable for the study or would prevent compliance with the study protocol

Note: Other protocol defined Inclusion/ Exclusion criteria may apply.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 187 (Actual)
Dates: Start 2015-04-30 (Actual); Primary Completion 2016-11-30 (Actual); Study Completion 2016-12-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Team, Study Director — Gilead Sciences
Locations (74):
- United States (33):
  - Digestive Health Specialists of The Southeast, Dothan, Alabama
  - Mayo Clinic, Scottsdale, Arizona
  - Cedars Sinai Medical Center, Los Angeles, California
  - South Denver Gastroenterology, Lone Tree, Colorado
  - University of Miami, Miami, Florida
  - Gastroenterology Group Of Naples, Naples, Florida
  - Gastroenterology Associates Of Central Georgia, LLC, Macon, Georgia
  - Medical Diagnostic Center (MDC)-Indiana University (IU) Health University Hospital, Indianapolis, Indiana
  - Iowa Digestive Disease Center, Clive, Iowa
  - Cotton-O'Neil Clinical Research Center, Digestive Health, Topeka, Kansas
  - Delta Research Partners, Monroe, Louisiana
  - Louisiana Research Center, Shreveport, Louisiana
  - University of Michigan, Ann Arbor, Michigan
  - Clinical Research Institute of Michigan, LLC, Chesterfield, Michigan
  - Mayo Clinic Rochester, Rochester, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - AGA Clinical Research Associates, LLC, Egg Harbor, New Jersey
  - Columbia University Medical Center/ New York Presbyterian, New York, New York
  - Premier Medical Group Of The Hudson Valley, Poughkeepsie, New York
  - Mayo Clinic Rochester, Rochester, New York
  - Asheville Gastroenterology Associates, Asheville, North Carolina
  - Consultants For Clinical Research, Cincinnati, Ohio
  - Great Lakes Gastroenterology, Mentor, Ohio
  - Gastro One, Germantown, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Texas Clinical Research Institute, Arlington, Texas
  - Ertan Digestive Disease Center of Excellence, UTH/MH-TMC, Houston, Texas
  - Gastroenterology Research of San Antonio, San Antonio, Texas
  - Gastroenterology Associates Of Tidewater, Chesapeake, Virginia
  - Digestive and Liver Disease Specialists, Norfolk, Virginia
  - Mcguire Dvamc, Richmond, Virginia
  - University of Washington Medical Center, Seattle, Washington
- Australia (5):
  - Concord Repatriation General Hospital, Concord, New South Wales
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Flinders Medical Centre, Bedford Park, South Australia
  - Footscray Hospital, Footscray, Victoria
  - Gastroenterology/Colorectal Medicine & Genetics, Melbourne, Victoria
- Canada (2):
  - Percuro Clinical Research Ltd., Victoria, British Columbia
  - Percuro Clinical Research Ltd., Victoria
- Czechia (2):
  - Hepato-Gastroenterologie Hk S.R.O., Hradec Králové
  - Ibd Clinical And Research Centre-Iscare Ivf, Prague
- France (4):
  - Hopital Beaujon, Clichy
  - CHRU de Lille, Lille
  - Chu Hotel Dieu-Chu De Nantes, Nantes
  - CHU de Saint Etienne - Hopital Nord, Saint-Priest-en-Jarez
- Germany (3):
  - Universitatsklinikum Schleswig-Holstein, Kiel
  - Eugastro Gmbh, Leipzig
  - Klinikum der Universitat Munchen, München
- Hungary (4):
  - Tolna Megye Balassa Janos Korhaz, Beri Balogh Adam
  - Rethy Pal Hospital-Clinic Bekescsaba, Békéscsaba
  - Pannonia Maganorvosi Centrum Kft, Budapest
  - Debreceni Egyeterm Orvos es Egeszsegtudomanyi Centrum, Debrecen
- Italy (2):
  - Universita Campus Biomedico, Roma
  - Humanitas Research Hospital, Rozzano
- New Zealand (3):
  - Christchurch Hospital, Christchurch
  - Southern District Health Board, Dunedin
  - Capital and Coast District Health board-Wellington hospital, Wellington
- Poland (7):
  - The Medical University of Bialystok Clinical, Bialystok
  - Gastromed, Lublin
  - Ai Centrum Medyczne, Poznan
  - CRC Sp. z o.o., Poznan
  - Endoskopia SP. z.o.o., Sopot
  - Centralny Szpital Kliniczny MSWiA, Warsaw
  - Lexmedica, Wroclaw
- South Africa (2):
  - Panorama Mediclinic Pvt Hospital, Panorama, Cape Town
  - Parklands Medical Centre, Durban
- Spain (4):
  - Hospital Universitari de Bellvitge, Barcelona
  - Hospital Universitario de Fuenlabrada, Fuenlabrada
  - Hospital Ramon y Cajal, Madrid
  - Hospital Universitari i Politecnic La Fe de Valencia, Valencia
- United Kingdom (3):
  - Norfolk and Norwich University Hospital Nhs Foundation Trust, Norwich, Norfolk
  - Cambridge University Hospitals NHS Foundation Trust, Cambridge
  - Oxford University Hospitals NHS Trust, Oxford

REFERENCES:
- [Result] Schreiber S, Siegel CA, Friedenberg KA, Younes ZH, Seidler U, Bhandari BR, Wang K, Wendt E, McKevitt M, Zhao S, Sundy JS, Lee SD, Loftus EV. A Phase 2, Randomized, Placebo-Controlled Study Evaluating Matrix Metalloproteinase-9 Inhibitor, Andecaliximab, in Patients With Moderately to Severely Active Crohn's Disease. J Crohns Colitis. 2018 Aug 29;12(9):1014-1020. doi: 10.1093/ecco-jcc/jjy070. PMID 29846530

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at study sites in North America, Europe, South Africa, and Asia Pacific. The first participant was screened on 30 April 2015. The last study visit occurred on 22 December 2016.
Pre-assignment Details: 315 participants were screened.
Groups:
- Andecaliximab 150 mg Every 2 Weeks: Double-Blind Phase: Participants received 1 single-use prefilled syringe (PFS) of andecaliximab 150 mg and matching placebo coadministered at Weeks 0, 2, 4, and 6 and 2 single-use PFS of placebo coadministered at Weeks 1, 3, 5 and 7.
  Open-Label Phase and Extended Treatment Phase: Participants received 1 single-use PFS of andecaliximab 150 mg administered weekly.
- Andecaliximab 150 mg Weekly: Double-Blind Phase: Participants received 1 single-use PFS of andecaliximab 150 mg and matching placebo coadministered weekly for 8 weeks.
  Open-Label Phase and Extended Treatment Phase: Participants received 1 single-use PFS of andecaliximab 150 mg administered weekly.
- Andecaliximab 300 mg Weekly: Double-Blind Phase: Participants received 2 single-use PFS of andecaliximab 150 mg coadministered weekly for 8 weeks.
  Open-Label Phase and Extended Treatment Phase: Participants received 1 single-use PFS of andecaliximab 150 mg administered weekly.
- Placebo: Double-Blind Phase: Participants received 2 single-use PFS of placebo coadministered weekly for 8 weeks.
  Open-Label and Extended Treatment Phase: Participants received 1 single-use PFS of andecaliximab 150 mg administered weekly.
Period: Double-Blind Phase (up to Week 8)
Arm/Group | Andecaliximab 150 mg Every 2 Weeks | Andecaliximab 150 mg Weekly | Andecaliximab 300 mg Weekly | Placebo
Started | 53 | 53 | 53 | 28
Completed | 52 | 48 | 47 | 27
Not Completed | 1 | 5 | 6 | 1
Not completed — Adverse Event | 0 | 2 | 4 | 1
Not completed — Withdrew Consent | 0 | 1 | 2 | 0
Not completed — Study Disease-Related Symptoms | 1 | 1 | 0 | 0
Not completed — Investigator's Discretion | 0 | 1 | 0 | 0
Period: Open-Label Phase (up to Week 52)
Arm/Group | Andecaliximab 150 mg Every 2 Weeks | Andecaliximab 150 mg Weekly | Andecaliximab 300 mg Weekly | Placebo
Started | 52 | 48 | 47 | 26 (1 participant completed Double-Blind Phase, but did not continue in Open-Label Phase.)
Completed | 4 | 3 | 2 | 2
Not Completed | 48 | 45 | 45 | 24
Not completed — Study Terminated by Sponsor | 27 | 28 | 28 | 13
Not completed — Investigator's Discretion | 14 | 11 | 11 | 2
Not completed — Adverse Event | 6 | 1 | 2 | 6
Not completed — Study Disease-Related Symptoms | 0 | 1 | 3 | 2
Not completed — Withdrew Consent | 1 | 2 | 1 | 1
Not completed — Lack of Efficacy | 0 | 1 | 0 | 0
Not completed — Lost to Follow-up | 0 | 1 | 0 | 0
Period: Extended Treatment Phase(up to Week 208)
Arm/Group | Andecaliximab 150 mg Every 2 Weeks | Andecaliximab 150 mg Weekly | Andecaliximab 300 mg Weekly | Placebo
Started | 3 (1 participant completed Open-Label Phase, but did not continue in Extended Treatment Phase.) | 2 (1 participant completed Open-Label Phase, but did not continue in Extended Treatment Phase.) | 2 | 2
Completed | 0 | 0 | 0 | 0
Not Completed | 3 | 2 | 2 | 2
Not completed — Study Terminated by Sponsor | 2 | 1 | 2 | 2
Not completed — Investigator's Discretion | 0 | 1 | 0 | 0
Not completed — Study Disease-Related Symptoms | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set included all participants who received at least 1 dose of study drug.
Groups:
- Andecaliximab 150 mg Every 2 Weeks: Double-Blind Phase: Participants received 1 single-use PFS of andecaliximab 150 mg and matching placebo coadministered at Weeks 0, 2, 4, and 6 and 2 single-use PFS of placebo coadministered at Weeks 1, 3, 5 and 7.
  Open-Label Phase and Extended Treatment Phase: Participants received 1 single-use PFS of andecaliximab 150 mg administered weekly.
- Total: Total of all reporting groups
Arm/Group | Andecaliximab 150 mg Every 2 Weeks | Andecaliximab 150 mg Weekly | Andecaliximab 300 mg Weekly | Placebo | Total
Number analyzed (Participants) | 53 | 53 | 53 | 28 | 187
Age, Continuous [Mean (Standard Deviation); unit: years] | 38 (12.8) | 39 (13.5) | 42 (11.7) | 38 (13.5) | 39 (12.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 28 | 22 | 15 | 90
  Male | 28 | 25 | 31 | 13 | 97
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: Asian | 1 | 1 | 0 | 1 | 3
  Race: Black or African American | 3 | 4 | 3 | 1 | 11
  Race: White | 48 | 42 | 48 | 22 | 160
  Race: Other | 1 | 0 | 1 | 3 | 5
  Race: Not Permitted | 0 | 6 | 1 | 1 | 8
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ethnicity: Hispanic or Latino | 1 | 1 | 5 | 1 | 8
  Ethnicity: Not Hispanic or Latino | 52 | 46 | 47 | 26 | 171
  Ethnicity: Not Permitted | 0 | 6 | 1 | 1 | 8
Region of Enrollment [Count of Participants; unit: Participants]
  Hungary | 2 | 1 | 0 | 2 | 5
  United States | 29 | 28 | 30 | 17 | 104
  Czechia | 1 | 2 | 1 | 1 | 5
  United Kingdom | 2 | 2 | 2 | 0 | 6
  Spain | 3 | 0 | 2 | 0 | 5
  New Zealand | 4 | 1 | 0 | 0 | 5
  Canada | 3 | 1 | 0 | 0 | 4
  Poland | 3 | 5 | 6 | 2 | 16
  Italy | 0 | 0 | 1 | 1 | 2
  South Africa | 0 | 0 | 2 | 1 | 3
  Australia | 3 | 2 | 3 | 1 | 9
  France | 0 | 6 | 1 | 1 | 8
  Germany | 3 | 5 | 5 | 2 | 15

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving Clinical Response (PRO2 Score ≤ 8) at Week 8 of the Double-Blind Phase
Description: Clinical response was defined as patient-reported outcomes (PRO2) score ≤ 8 at Week 8. PRO2 is the weighted average of the 2 variables of frequency of liquid or very soft stool and abdominal pain, based on 7-day participant diary data. The PRO2 score has a minimum score of 0 and has no upper bound, with a higher score indicating more frequent stools and more severe abdominal pain. Week 8 refers to the analysis window of Day 43 to Day 70 and prior to the first Open-Label dose date. Participants with a missing PRO2 value at the Week 8 analysis visit were imputed as not achieving the Clinical Response.
Time Frame: Week 8
Population: Full Analysis Set included all randomized participants who received at least 1 dose of study drug.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Andecaliximab 150 mg Every 2 Weeks | Andecaliximab 150 mg Weekly | Andecaliximab 300 mg Weekly | Placebo
Number analyzed (Participants) | 53 | 53 | 53 | 28
percentage of participants | 17.0 [8.1 to 29.8] | 13.2 [5.5 to 25.3] | 11.3 [4.3 to 23.0] | 14.3 [4.0 to 32.7]

2. Primary Outcome: Percentage of Participants Achieving Endoscopic Response (≥ 50% Reduction From Baseline SES-CD) at Week 8 of the Double-Blind Phase
Description: Endoscopic response was defined as ≥ 50% reduction from baseline in Simple Endoscopic Score for Crohn's Disease (SES-CD) at Week 8. The SES-CD evaluates 4 endoscopic variables: ulcer size, ulcerated surface, affected surface, and presence of narrowings. The total SES-CD is calculated as the sum of the 4 variables for the 5 bowel segments: rectum, left colon, transverse colon, right colon, and ileum. Scores range from 0 to 60, with higher scores indicating more severe disease. Week 8 refers to the analysis window of Day 43 to Day 70 and prior to the first Open-Label dose date. Participants with missing SES-CD value at Week 8 analysis visit were imputed as not achieving Endoscopic Response.
Time Frame: Week 8
Population: Participants in the Full Analysis Set were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Andecaliximab 150 mg Every 2 Weeks | Andecaliximab 150 mg Weekly | Andecaliximab 300 mg Weekly | Placebo
Number analyzed (Participants) | 53 | 53 | 53 | 28
percentage of participants | 11.3 [4.3 to 23.0] | 13.2 [5.5 to 25.3] | 7.5 [2.1 to 18.2] | 10.7 [2.3 to 28.2]

3. Secondary Outcome: Percentage of Participants Achieving CDAI Remission (CDAI ≤ 150) at Week 8 of the Double-Blind Phase
Description: Clinical remission was defined as Crohn's Disease Activity Index (CDAI) ≤ 150 at Week 8. CDAI is used as a measure of clinical response and remission. It includes 8 variables of patient-reported symptoms and objective variables: stool count, abdominal pain, general well-being, complications, use of anti-diarrheal medications, presence of abdominal mass, hematocrit values, and weight. It has a minimum range of 0 and no upper bound, with higher scores indicating greater disease activity. Week 8 refers to the analysis window of Day 43 to Day 70 and prior to the first Open-Label dose date. Participants with missing CDAI score at Week 8 analysis visit were imputed as not achieving CDAI Remission.
Time Frame: Week 8
Population: Participants in the Full Analysis Set were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Andecaliximab 150 mg Every 2 Weeks | Andecaliximab 150 mg Weekly | Andecaliximab 300 mg Weekly | Placebo
Number analyzed (Participants) | 53 | 53 | 53 | 28
percentage of participants | 20.8 [10.8 to 34.1] | 17.0 [8.1 to 29.8] | 11.3 [4.3 to 23.0] | 21.4 [8.3 to 41.0]

4. Secondary Outcome: Percentage of Participants Achieving Mucosal Healing (SES-CD Size-of-Ulcer Subscore = 0) at Week 8 of the Double-Blind Phase
Description: The SES-CD evaluates 4 endoscopic variables: ulcer size, ulcerated surface, affected surface, and presence of narrowings. The SES-CD size-of-ulcer subscore ranges from 0 (none) to 3 (very large). Mucosal healing at Week 8 was defined as the size-of-ulcer subscore for segments with non-zero baseline value changes to zero at Week 8 AND the size-of-ulcer subscore for segments with zero value at baseline remain zero at Week 8. Week 8 refers to the analysis window of Day 43 to Day 70 and prior to the first Open-Label dose date. Participants with missing SES-CD size-of-ulcer subscore at Week 8 analysis visit were imputed as not achieving Mucosal Healing.
Time Frame: Week 8
Population: Participants in the Full Analysis Set were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Andecaliximab 150 mg Every 2 Weeks | Andecaliximab 150 mg Weekly | Andecaliximab 300 mg Weekly | Placebo
Number analyzed (Participants) | 53 | 53 | 53 | 28
percentage of participants | 5.7 [1.2 to 15.7] | 1.9 [0.0 to 10.1] | 1.9 [0.0 to 10.1] | 7.1 [0.9 to 23.5]

ADVERSE EVENTS:
Time Frame: Double-Blind Phase: First dose of andecaliximab to Week 8; Open-Label Phase (includes adverse events occurring in the Extended Treatment Phase): First dose of open label andecaliximab to the last dose date (maximum: 200 weeks) plus 30 days
Description: Safety Analysis Set (Double-Blind Phase and Open-Label Phase) included all participants who received at least 1 dose of study drug.
Groups:
- Double-Blind Andecaliximab 150 mg Every 2 Weeks (Q2W): Adverse events reported in this group occurred during the Double-Blind Phase. Participants received 1 single-use PFS of andecaliximab 150 mg and matching placebo coadministered at Weeks 0, 2, 4, and 6 and 1 single-use PFS of placebo coadministered at Weeks 1, 3, 5 and 7.
- Double-Blind Andecaliximab 150 mg Weekly (QW): Adverse events reported in this group occurred during the Double-Blind Phase. Participants received 1 single-use PFS of andecaliximab 150 mg and matching placebo coadministered weekly for 8 weeks.
- Double-Blind Andecaliximab 300 mg Weekly: Adverse events reported in this group occurred during the Double-Blind Phase. Participants received 2 single-use PFS of andecaliximab 150 mg coadministered weekly for 8 weeks.
- Double-Blind Placebo: Adverse events reported in this group occurred during the Double-Blind Phase. Participants received 2 single-use PFS of placebo coadministered weekly for 8 weeks.
- Open-Label Andecaliximab QW From Andecaliximab 150 mg Q2W: Adverse events reported in this group occurred during the Open-Label Phase in participants who received andecaliximab 150 mg weekly after switching from the Double-Blind Andecaliximab 150 mg Every 2 Weeks group.
- Open-Label Andecaliximab QW From Andecaliximab 150 mg QW: Adverse events reported in this group occurred during the Open-Label Phase in participants who received andecaliximab 150 mg weekly after switching from the Double-Blind Andecaliximab 150 mg Weekly group.
- Open-Label Andecaliximab QW From Andecaliximab 300 mg QW: Adverse events reported in this group occurred during the Open-Label Phase in participants who received andecaliximab 150 mg weekly after switching from the Double-Blind Andecaliximab 300 mg Every 2 Weeks group.
- Open-Label Andecaliximab QW From Placebo: Adverse events reported in this group occurred during the Open-Label Phase in participants who received andecaliximab 150 mg weekly after switching from the Double-Blind Placebo group.
Arm/Group | Double-Blind Andecaliximab 150 mg Every 2 Weeks (Q2W) | Double-Blind Andecaliximab 150 mg Weekly (QW) | Double-Blind Andecaliximab 300 mg Weekly | Double-Blind Placebo | Open-Label Andecaliximab QW From Andecaliximab 150 mg Q2W | Open-Label Andecaliximab QW From Andecaliximab 150 mg QW | Open-Label Andecaliximab QW From Andecaliximab 300 mg QW | Open-Label Andecaliximab QW From Placebo
All-Cause Mortality (participants affected / at risk) | 0/53 | 0/53 | 0/53 | 0/28 | 0/52 | 0/48 | 0/47 | 0/26
Serious Adverse Events (participants affected / at risk) | 1/53 | 6/53 | 8/53 | 3/28 | 9/52 | 10/48 | 7/47 | 6/26
Other Adverse Events (participants affected / at risk) | 15/53 | 25/53 | 25/53 | 13/28 | 22/52 | 21/48 | 17/47 | 16/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Double-Blind Andecaliximab 150 mg Every 2 Weeks (Q2W) (N=53) | Double-Blind Andecaliximab 150 mg Weekly (QW) (N=53) | Double-Blind Andecaliximab 300 mg Weekly (N=53) | Double-Blind Placebo (N=28) | Open-Label Andecaliximab QW From Andecaliximab 150 mg Q2W (N=52) | Open-Label Andecaliximab QW From Andecaliximab 150 mg QW (N=48) | Open-Label Andecaliximab QW From Andecaliximab 300 mg QW (N=47) | Open-Label Andecaliximab QW From Placebo (N=26)
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0
Anal fistula (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Crohn's disease (Gastrointestinal disorders) | 0 | 3 | 2 | 0 | 4 | 5 | 4 | 3
Fistula of small intestine (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Ileal stenosis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Intestinal perforation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Large intestinal stenosis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Large intestine perforation (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Proctalgia (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 2 | 1 | 2 | 0
Abdominal abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Anal abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Appendicitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Bacterial pyelonephritis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Clostridium difficile infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Cytomegalovirus infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Enteritis infectious (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Perirectal abscess (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Post procedural complication (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Post procedural haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Procedural pain (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Acute prerenal failure (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Acne (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Peripheral ischaemia (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Double-Blind Andecaliximab 150 mg Every 2 Weeks (Q2W) (N=53) | Double-Blind Andecaliximab 150 mg Weekly (QW) (N=53) | Double-Blind Andecaliximab 300 mg Weekly (N=53) | Double-Blind Placebo (N=28) | Open-Label Andecaliximab QW From Andecaliximab 150 mg Q2W (N=52) | Open-Label Andecaliximab QW From Andecaliximab 150 mg QW (N=48) | Open-Label Andecaliximab QW From Andecaliximab 300 mg QW (N=47) | Open-Label Andecaliximab QW From Placebo (N=26)
Anaemia (Blood and lymphatic system disorders) | 0 | 2 | 6 | 0 | 1 | 1 | 1 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 7 | 4 | 3 | 7 | 1 | 3 | 1
Crohn's disease (Gastrointestinal disorders) | 1 | 1 | 2 | 2 | 6 | 10 | 4 | 5
Nausea (Gastrointestinal disorders) | 3 | 1 | 7 | 5 | 3 | 4 | 1 | 2
Vomiting (Gastrointestinal disorders) | 2 | 1 | 1 | 1 | 3 | 0 | 2 | 0
Fatigue (General disorders) | 6 | 0 | 5 | 1 | 1 | 1 | 0 | 0
Pyrexia (General disorders) | 1 | 3 | 0 | 4 | 2 | 1 | 2 | 2
Clostridium difficile infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2
Herpes zoster (Infections and infestations) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 2 | 1 | 4 | 0 | 4 | 3 | 4 | 1
Rhinitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 1 | 2 | 1 | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 1 | 2 | 1 | 1 | 0 | 3 | 1 | 1
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0
Hepatic enzyme increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 3 | 4 | 1 | 2 | 2 | 1 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 4 | 1 | 2 | 2 | 0 | 1 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 2 | 0 | 2 | 0 | 1 | 0 | 1
Dizziness (Nervous system disorders) | 0 | 5 | 2 | 0 | 0 | 0 | 1 | 0
Headache (Nervous system disorders) | 0 | 4 | 5 | 1 | 2 | 1 | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 1 | 2 | 2 | 1 | 0 | 0

LIMITATIONS AND CAVEATS:
A prespecified topline analysis was performed after the last enrolled subject received the 8-week Double-Blind induction treatment. Based on this review, Gilead terminated the Open-Label and Extended Treatment Phases of study due to lack of efficacy.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years